CLINICAL TRIAL: NCT06842017
Title: Passive Exoskeletons for Supporting Patients With Shoulder Musculoskeletal Disorders in Daily Activities: Assessment of Impact and User Experience
Brief Title: Passive Exoskeletons for Assisting Patients With Shoulder Musculoskeletal Disorders
Acronym: EXOADL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Umile Giuseppe Longo, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 271.24 CET2PUDcbm; PNC0000007 - CUP: B53C22006980 (Other Grant/Funding Number: Italian Ministry of Research, under the complementary actions to the NRRP "Fit4MedRob - Fit for Medical Robotics")
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Musculoskeletal Disorders
Keywords: Musculoskeletal disorders; Shoulder rehabilitation; Exoskeletons; Pain management; Assistive technology; Patient outcomes; Biomechanics
MeSH Terms: conditions — Musculoskeletal Diseases; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with shoulder musculoskeletal disorders (Experimental): The study will involve 15 adults with shoulder musculoskeletal disorders. Eligible participants must be over 18 years old and diagnosed with conditions such as rotator cuff tears, adhesive capsulitis, or osteoarthritis. Individuals with neurological conditions, infections, inflammatory diseases, prior major shoulder surgeries, or those who are pregnant will be excluded. After obtaining informed consent, baseline demographic and anthropometric data will be collected. Patients will be assessed during a series of experimental sessions at the Lab of Motion Analysis, where they will perform relevant activities of daily living (ADLs) with and without the assistance of a passive exoskeleton. These sessions will include evaluations of joint functionality, pain, and muscle activity using wearable sensors, EMG measurements, and kinematic analysis.
  Interventions: Device: Passive Exoskeleton.; Procedure: Shoulder Rehabilitation with Passive Exoskeleton.; Other: Usability Assessment and Patient Satisfaction.

INTERVENTIONS:
Device: Passive Exoskeleton. — The passive exoskeleton is used to assist patients with shoulder musculoskeletal disorders during the performance of activities of daily living (ADLs), such as overhead reaching and lifting. The device helps reduce biomechanical load and muscle strain, providing support for the shoulder joint.
Procedure: Shoulder Rehabilitation with Passive Exoskeleton. — The rehabilitation protocol involves the use of a passive exoskeleton during physical tasks to improve shoulder function and reduce pain. Patients perform specific exercises while wearing the exoskeleton, which is tailored to their individual needs.
Other: Usability Assessment and Patient Satisfaction. — The usability of the passive exoskeleton is evaluated using validated scales, such as the System Usability Scale (SUS), to assess its comfort, effectiveness, and overall satisfaction. The assessment also includes patient feedback on the ease of use and perceived benefits of the device during rehabilitation sessions.

SUMMARY:
Goal: The clinical investigation aims to evaluate the usability of passive exoskeletons, their impact on daily living activities, and the perceived experience of patients with shoulder musculoskeletal disorders. This will be assessed through specific validated questionnaires.

Participant Population: The study will enroll 15 participants diagnosed with shoulder musculoskeletal disorders, including rotator cuff tears, adhesive capsulitis, and glenohumeral osteoarthritis. Participants must be employed in physically demanding jobs that require frequent upper limb activity.

Main Questions:

* How does the integration of passive exoskeletons in daily activities influence usability and functional performance in patients with shoulder musculoskeletal disorders?
* To what extent does the use of passive exoskeletons improve the perceived physical effort and quality of life in these patients?
* How do patients perceive the comfort and effectiveness of passive exoskeletons during the execution of daily living tasks?

Participant Tasks:

* Comprehensive shoulder physical examination. Instruction on the proper use of the Paexo passive exoskeleton and customization of its settings.
* Execution of workplace-relevant tasks (e.g., lifting, overhead reaching) with and without the exoskeleton.
* Evaluation of usability, comfort, and perceived workload using validated scales such as the System Usability Scale (SUS), NASA Task Load Index (NASA-TLX), and Technology Acceptance Model (TAM).

DETAILED DESCRIPTION:
Shoulder musculoskeletal disorders, such as rotator cuff injuries, adhesive capsulitis, and osteoarthritis, severely impact daily activities due to pain, reduced mobility, and muscle weakness. These conditions limit tasks like lifting, reaching, and even simple activities such as dressing or combing hair, significantly affecting patients' quality of life. While traditional physiotherapy can help, barriers such as limited access and poor adherence to home exercises hinder its effectiveness. This has led to the exploration of new rehabilitation methods, particularly passive exoskeletons.

Passive exoskeletons, which use mechanical components like springs to assist movement without external power, have shown potential in reducing muscle strain and supporting tasks requiring arm elevation or lifting. These devices are lightweight, cost-effective, and easy to use, but research on their application for patients with musculoskeletal disorders is limited.

This study aims to assess the impact of passive exoskeletons on joint functionality, pain reduction, and performance of activities of daily living (ADLs) in patients with shoulder disorders. It will also evaluate the usability and comfort of the devices using validated questionnaires. Participants will be enrolled from the FPUCBM Unit of Traumatology and Sports Medicine and undergo experimental sessions involving movement tasks with and without the exoskeleton. The study will measure biomechanical effects, pain levels, and user satisfaction, with the ultimate goal of integrating passive exoskeletons into clinical rehabilitation protocols to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age over 18 years.
* Employment in a physically demanding job requiring frequent upper limb activity.
* Diagnosis of one of the following conditions related to shoulder musculoskeletal disorders: rotator cuff tears, massive tears with pseudoparalytic limb, adhesive capsulitis, post-surgical outcomes following rotator cuff repair or reverse shoulder arthroplasty, and glenohumeral osteoarthritis.
* Signed informed consent.

Exclusion Criteria

* Failure to provide signed informed consent.
* Any condition that hinders the use of exoskeletons.
* Insufficient cognitive or language abilities to follow instructions provided by clinicians and/or investigators.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of Joint Range of Motion (ROM) | a single session up to one year from the subject's enrollment
  Joint Range of Motion (ROM) will be evaluated using stereophotogrammetric systems, and wearable sensors during the execution of movements with and without the exoskeleton
Pain Assessment using the Visual Analogue Scale (VAS) before and after exoskeleton use | a single session up to one year from the subject's enrollment, before and after exoskeleton use
  Pain levels will be measured using the Visual Analogue Scale (VAS) before and after exoskeleton use. The VAS provides a quantitative measure of pain intensity, with scores ranging from 0 (no pain) to 10 (worst pain imaginable).
Evaluation of the American Shoulder and Elbow Surgeons Score (ASES) | a single session up to one year from the subject's enrollment
  The ASES score will be used to evaluate shoulder function and pain. This clinical scale assesses both pain and the ability to perform daily activities, with higher scores indicating better function. The total score ranges from 0 to 100, with 0 representing the worst shoulder function and 100 indicating the best possible outcome.
Evaluation of the Disabilities of the Arm, Shoulder, and Hand Score (DASH) | a single session up to one year from the subject's enrollment
  The DASH questionnaire will assess disability and symptoms in people with upper limb musculoskeletal disorders. Higher scores indicate greater disability. The total score ranges from 0 to 100, with 0 representing no disability and 100 indicating the most severe disability.
Evaluation of the Short Form Health Survey 36 (SF-36) | a single session up to one year from the subject's enrollment
  The SF-36 will evaluate overall health-related quality of life, covering physical functioning, bodily pain, and general health perceptions. Higher scores indicate better health status. The total score ranges from 0 to 100, with 0 representing the poorest health status and 100 indicating the best possible health status.
Evaluation of the Shoulder Pain and Disability Index (SPADI) | a single session up to one year from the subject's enrollment
  The SPADI will measure pain and disability associated with shoulder pathology. It consists of two subscales: pain and disability, with higher scores indicating greater impairment. The total score ranges from 0 to 100, with 0 representing no impairment and 100 indicating the most severe impairment.
Heart Rate evaluation with and without the exoskeleton | a single session up to one year from the subject's enrollment
  Heart rate will be monitored using wearable sensors during tasks performed with and without the exoskeleton. The heart rate will be recorded in beats per minute to evaluate the physiological response to movement efficiency and task execution.
Electromyographic Activity (EMG) evaluation with and without the exoskeleton | a single session up to one year from the subject's enrollment
  Muscle activity in key shoulder muscles, such as the anterior deltoid and upper trapezius, will be measured using electromyographic (EMG) sensors during movement execution with and without the exoskeleton. The EMG signal will be recorded in millivolts (mV) to quantify the level of muscle activation and the physiological response during movement execution.
Respiratory Rate Evaluation with and without exoskeleton | A single session up to one year from the subject's enrollment
  Respiratory rate will be monitored using wearable sensors during tasks performed with and without the exoskeleton. The respiratory rate will be recorded in breaths per minute to assess the physiological response and efficiency of breathing during movement execution.

SECONDARY OUTCOMES:
Evaluation of the Usability Level of the passive exoskeleton using the System Usability Scale (SUS) | a single session up to one year from the subject's enrollment
  The usability of the passive exoskeleton will be assessed using the System Usability Scale (SUS), a standardized questionnaire consisting of ten statements rated on a five-point Likert scale from "Strongly Disagree" to "Strongly Agree." Higher scores indicate better usability.
Evaluation of the Patient satisfaction with the exoskeleton using the Technology Acceptance Model (TAM) | a single session up to one year from the subject's enrollment
  Patient satisfaction with the exoskeleton will be measured using the Technology Acceptance Model (TAM), which evaluates technology acceptability and usability, focusing on perceived ease of use and usefulness. Scores range from 0 to 100, with higher scores indicating greater acceptance and usability.
Assessment of Patient-Perceived Workload Using the NASA Task Load Index (NASA-TLX) | a single session up to one year from the subject's enrollment
  Patient workload will be assessed using the NASA Task Load Index (NASA-TLX), which evaluates perceived workload across several dimensions, including mental demand, physical demand, temporal demand, performance, effort, and frustration. Scores range from 0 to 100, with higher scores indicating a greater perceived workload.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The ownership of the data is of the promoter and shared with the investigators and will be managed according to the agreements between the participating institutions and with the researchers. Data Property belongs to Fondazione Policlinico Universitario Campus Bio-Medico. The personnel involved in this study will have access to all data. In agreement with the ICH-GCP, the principal investigator of the study agrees to produce a report on the study, share all the data collected as described in the Protocol, and ensure that the data are reported responsibly and consistently.
  The transmission or dissemination of data through scientific publications and/or presentations in congresses, conferences, seminars, and participation in multicenter studies will take place exclusively following a purely statistical processing of the same, or in any case, in an anonymous form.